CLINICAL TRIAL: NCT06013306
Title: Long-Term Follow-up Study of Subjects With Knee Osteoarthritis Who Had Administered FURESTEM-OA Kit Inj. in K0701 Study
Status: Not yet recruiting | Type: Observational
Sponsor: Kang Stem Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: K0701-E
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Long-Term Follow-up Study of Subjects with Knee Osteoarthritis who had administered FURESTEM-OA Kit Inj. in K0701 study

ELIGIBILITY:
Inclusion Criteria:

* Those who participated in the K0701 clinical trial and received PureStem-OA Kit Inj
* Those who understand and voluntarily sign an informed consent form

exclusion criteria

* None

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those who participated in the K0701 clinical trial and received PureStem-OA Kit Inj
Sampling Method: Non-Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2023-09-14 (Estimated); Primary Completion 2029-11-07 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of AESI | 5 years follow-up after treatment
Number of SS | 5 years follow-up after treatment

SECONDARY OUTCOMES:
Changes in Knee Injury and Osteoarthritis Outcome Score (KOOS) | 1 year (52 weeks), 2 years (104 weeks), and 3 years (156 weeks) after treatment
  The higher the score, the worse the condition of the disease is.
Changes in Western Ontario and McMaster Universities osteoarthritis index (WOMAC) | 1 year (52 weeks), 2 years (104 weeks), and 3 years (156 weeks) after treatment
  The WOMAC evaluation is evaluated using the score value converted through the KOOS evaluation paper.
Changes in 100-mm VAS | 1 year (52 weeks), 2 years (104 weeks), and 3 years (156 weeks) after treatment
Changes in International Knee Documentation Committee Scoring System (IKDC) | 1 year (52 weeks), 2 years (104 weeks), and 3 years (156 weeks) after treatment
  A higher score indicates better function and less symptomatic
Evaluation of International K&L grade(X-ray) | 1 year (52 weeks), 2 years (104 weeks), and 3 years (156 weeks) after treatment
  Grade 0 - No radioligical findings of osteoarthritis Grade 1 - Doubtful narrowing of joint space and possible osteophytic lipping Grade 2 - Definite osteophytes and possible narrowing of joint space Grade 3 - Moderate osteophytes, definite narrowing of joint space, and some sclerosis and deformity of bone ends Grade 4 - Large osteophytes, marked narrowing of joint space, severe sclerosis, and definite deformity of bone ends
Magnetic Resonance Observation of Cartilage Repair Tissue (MOCART) scores(MRI) | 1 year (52 weeks), 2 years (104 weeks), and 3 years (156 weeks) after treatment
  A higher score indicates better function and less symptomatic
Whole-Organ Magnetic Resonance Imaging Score (WORMS) score | 1 year (52 weeks), 2 years (104 weeks), and 3 years (156 weeks) after treatment
  The higher the score means normal state.

CONTACTS AND LOCATIONS:
Overall Officials: Kyoung-Ho Yoon, professor (CI), Principal Investigator — Kyung Hee University Hospital; Sang Hak Lee, professor, Principal Investigator — Gangdong Kyunghee University Hospital